CLINICAL TRIAL: NCT06354660
Title: A Phase 3, Randomized, Multicenter, Double-Blind Study to Investigate the Efficacy and Safety of Retatrutide Once Weekly Compared With Placebo in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise Alone (TRANSCEND-T2D-1)
Brief Title: Effect of Retatrutide Compared With Placebo in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise Alone (TRANSCEND-T2D-1)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18804; J1I-MC-GZBY (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Type 2
Keywords: Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Retatrutide Dose Level 1 (Experimental): Participants will receive retatrutide administered subcutaneously (SC).
  Interventions: Drug: Retatrutide
- Retatrutide Dose Level 2 (Experimental): Participants will receive retatrutide administered SC.
  Interventions: Drug: Retatrutide
- Retatrutide Dose Level 3 (Experimental): Participants will receive retatrutide administered SC.
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC.
  Other Names: LY3437943
  Arms: Retatrutide Dose Level 1; Retatrutide Dose Level 2; Retatrutide Dose Level 3
Drug: Placebo — Administered SC.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of retatrutide compared with placebo in participants with Type 2 Diabetes and inadequate glycemic control. The study will last about 11 months and may include up to 11 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes (T2D)
* Have HbA1c ≥ 7.0% to ≤ 9.5%
* Are naïve to insulin therapy and have not used oral or injectable antihyperglycemic (diabetes) medication for at least 90 days prior to screening
* Are of stable weight for at least 90 days prior to screening
* Have a Body Mass Index (BMI) ≥ 23.0 kilograms per meter squared (kg/m^2)

Exclusion Criteria:

* Have Type 1 Diabetes (T1D)
* Have a history of ketoacidosis or hyperosmolar state or coma within the last 6 months prior to screening
* Have a history of severe hypoglycemia or hypoglycemia unawareness within the last 6 months prior to screening
* Are currently receiving or planning to receive treatment for diabetic retinopathy and/or macular edema
* Have an estimated glomerular filtration rate (eGFR) <15 milliliters/minute/1.73 meter squared (mL/min/1.73 m^2) as determined by the central laboratory
* Have a prior or planned surgical treatment for obesity
* Have New York Heart Association Functional Classification IV congestive heart failure
* Have had an acute myocardial infarction, stroke, or were hospitalized for congestive heart failure within 90 days prior to screening
* Have a known clinically significant gastric emptying abnormality
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years
* Have any lifetime history of a suicide attempt
* Had chronic or acute pancreatitis
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) syndrome Type 2
* Have taken prescribed or over-the-counter medication, or alternative remedies, intended to promote body weight reduction within 90 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) (%) | Baseline, Week 40

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve HbA1c < 7.0% | Week 40
Percentage of Participants Who Achieve HbA1c ≤ 6.5% | Week 40
Percentage of Participants Who Achieve HbA1c < 5.7% | Week 40
Change from Baseline in Fasting Serum Glucose | Baseline, Week 40
Percent Change from Baseline in Body Weight | Baseline, Week 40
Change from Baseline in Body Weight | Baseline, Week 40
Percentage of Participants Who Achieve Weight Reduction of ≥ 5% | Week 40
Percentage of Participants Who Achieve Weight Reduction of ≥ 10% | Week 40
Percentage of Participants Who Achieve Weight Reduction of ≥ 15% | Week 40
Percentage of Participants Who Achieve HbA1c ≤ 6.5% and ≥ 10% Weight Reduction | Week 40
Percent Change from Baseline in Triglycerides | Baseline, Week 40
Percent Change from Baseline in Non- High-Density Lipoprotein (HDL) Cholesterol | Baseline, Week 40
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 40

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (48):
- United States (29):
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Tucson Clinical Research Institute, Tucson, Arizona
  - San Fernando Valley Health Institute, Canoga Park, California
  - Ark Clinical Research, Long Beach, California
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - New Horizon Research Center, Miami, Florida
  - Ezy Medical Research, Miami, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Trinity Research Centers, Marietta, Georgia
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Clinical Research Professionals, Chesterfield, Missouri
  - Boeson Research MSO, Missoula, Montana
  - NJ MedCare & NJ Heart, Linden, New Jersey
  - Accellacare - Wilmington - 1917 Tradd Court, Wilmington, North Carolina
  - Providence Health Partners-Center for Clinical Research, Dayton, Ohio
  - Clinical Research of Philadelphia, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Delricht Research - Tobias Gadson Boulevard - Charleston, Charleston, South Carolina
  - Lifedoc Research - Lenox Park Drive, Memphis, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Prime Revival Research Institute, LLC, Flower Mound, Texas
  - Valley Institute of Research - Fort Worth, Fort Worth, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - MultiCare Rockwood Cheney Clinic, Cheney, Washington
  - Eastside Research Associates, Redmond, Washington
- India (8):
  - All India Institute of Medical Sciences, Raipur, Chhattisgarh
  - Gujarat Endocrin Pvt Ltd, Ahmedabad, Gujarat
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - Victoria Hospital, Bangalore Medical College And Research Institute, Bangalore, Karnataka
  - Government Medical College - Kozhikode, Kozhikode, Kerala
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Eternal Heart Care Center and Research Institute, Jaipur, Rajasthan
  - Brij Medical Centre Private Limited, Kanpur, Uttar Pradesh
- Mexico (9):
  - Grupo Ollin Care, Pachuca, Hidalgo
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad, Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Unidad biomedica avanzada monterrey, Monterrey, Nuevo León
  - Clínica García Flores SC, Monterrey, Nuevo León
  - Centro de investigación y control metabólico, San Nicolás de los Garza, Nuevo León
  - EME RED Hospitalaria, Mérida, Yucatán
  - Medical Care and Research SA de CV, Mérida, Yucatán
  - Arké SMO S.A de C.V, Veracruz
- Puerto Rico (2):
  - Dorado Medical Complex, Dorado
  - Ponce Medical School Foundation Inc., Ponce

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Effect of Retatrutide Compared With Placebo in Adult Participants With Type 2 Diabetes and Inadequate Glycemic Control With Diet and Exercise Alone (TRANSCEND-T2D-1) — https://trials.lilly.com/en-US/trial/472275